CLINICAL TRIAL: NCT00267345
Title: Measurement of Hormonal Concentration in Chylothorax Fluid in Infants With Congenital Chylothorax
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Other Study IDs: SHEBA-05-3927-JK-CTIL
Record Dates: First submitted 2005-12-19; First posted 2005-12-20 (Estimated); Last update posted 2007-03-01 (Estimated); Status verified 2006-01

CONDITIONS: Congenital Chylothorax
MeSH Terms: conditions — Chylothorax, congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Late onset Hypothyroidism was found in infant with congenital hypothyroidism. The hypothesis is that infants with congenital hypothyroidism may lose thyroxin and other hormones via the chylothorax fluid causing transient hypothyroidism. In this study hormonal concentration will be measured in the chyle as well as hormonal serum level.

DETAILED DESCRIPTION:
Late onset Hypothyroidism was found in infant with congenital hypothyroidism. The hypothesis is that infants with congenital hypothyroidism may lose thyroxin and other hormones via the chylothorax fluid causing transient hypothyroidism. In this study hormonal concentration will be measured in the chyle as well as hormonal serum level.

ELIGIBILITY:
Inclusion Criteria:

* Infants with congenital chylothorax requiring thorax drain

Exclusion Criteria:

* none

Ages: 1 Hour to 10 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15
Dates: Start 2005-03; Study Completion 2007-10

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Kuint, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel